CLINICAL TRIAL: NCT04164056
Title: Hippocampal and Thalamic Deep Brain Stimulation for Bilateral Temporal Lobe Epilepsy
Brief Title: Hippocampal and Thalamic DBS for Bilateral Temporal Lobe Epilepsy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Beijing Tiantan Hospital (Other); The Second Hospital of Hebei Medical University (Other); Zhejiang Provincial People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-192
Record Dates: First submitted 2019-10-10; First posted 2019-11-15 (Actual); Last update posted 2019-11-15 (Actual); Status verified 2019-10

CONDITIONS: Epilepsy, Temporal Lobe
MeSH Terms: conditions — Epilepsy, Temporal Lobe | interventions — Deep Brain Stimulation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- stimulation on the hippocampus (Experimental): deep brain stimulation on the hippocampus
  Interventions: Device: deep brain stimulation
- stimulation on the anterior nucleus of the thalamus (Active Comparator): deep brain stimulation on the anterior nucleus of the thalamus
  Interventions: Device: deep brain stimulation

INTERVENTIONS:
Device: deep brain stimulation — deep brain stimulation on the hippocampus or the anterior nucleus of the thalamus

SUMMARY:
The study aims to compare the safety and effectiveness of deep brain stimulation of the hippocampus and the anterior nucleus of the thalamus for reducing the frequency of seizures in patients with bilateral temporal lobe epilepsy.

DETAILED DESCRIPTION:
The outcome of resective surgery for bilateral temporal lobe epilepsy (BTLE) is poor. Neuromodulation such as deep brain stimulation is an alternative therapy for patients with drug-resistant epilepsy, especially for those not suitable for resective surgery. This prospective, randomized, open-label trial aims to compare the effectiveness of deep brain stimulation of the hippocampus and the anterior nucleus of the thalamus for bilateral temporal lobe epilepsy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients between 12 to 60 years old.
2. Bilateral temporal lobe epilepsy patients proved by VEEG or SEEG.
3. At least 3 seizures per month but not more than 10 seizures per month, and the longest seizure interval is no more than 30 days during the baseline.
4. Patients failed to at least 3 antiepileptic drugs (AEDs), and are receiving at least 1 AEDs now.
5. Be able to complete seizure diary.
6. Agree to participate this study and sign informed consent.

Exclusion Criteria:

1. Extratemporal lobe epilepsy or with potential extratemporal epileptogenic focus.
2. Patients with psychogenic non-epileptic seizures.
3. IQ < 70, or unable to complete the study.
4. Patients are pregnant or plan for it.
5. Patients with implanted electrical stimulation medical device.
6. Patients with other severe neuropsychiatric disorders such as dementia, schizophrenia, or neurodegenerative diseases.
7. Patients with cerebral lesions which unsuitable for lead implantation.

Ages: 12 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-11 (Estimated); Primary Completion 2022-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Responder Rate | 3 years after DBS
  The rate of patients response to DBS, patients have at least 50% decrease in average seizure frequency after DBS are considered as responder.
Seizure-Free Rate | 3 years after DBS
  The rate of patients who achieve seizure free after DBS. Patients don't have seizure for at least 1 year are considered seizure free.
Change in Seizure Frequency | 3 years after DBS
  The seizure frequency after DBS compared to the seizure frequency in baseline.

SECONDARY OUTCOMES:
Change in Percentage of Seizure-free Days | 1 year and 3 years after DBS
  The percentage of seizure-free days after DBS compared to the percentage of seizure-free days in baseline.
Change in the Maximum Length of Seizure Intervals | 1 year and 3 years after DBS
  The maximum length of seizure intervals after DBS compared to the maximum length of seizure intervals in baseline.
Change in GTCS Frequency | 1 year and 3 years after DBS
  The GTCS frequency after DBS compared to the GTCS frequency in baseline.
Incidence Rate of Sudden Unexplained Death in Epilepsy (SUDEP) | 1 year and 3 years after DBS
  The Incidence Rate after DBS.
Change in Memory | 1 year and 3 years after DBS
  The memory test scores after DBS compared to baseline. Wechsler memory scale (WMS, ≤51 ~ 150, higher scores mean better outcome)
Change in Cognitive Function | 1 year and 3 years after DBS
  The cognitive test scores after DBS compared to baseline. Montreal Cognitive Assessment(MoCA, 0-30 scores, higher scores mean better outcome)
Change in Depression | 1 year and 3 years after DBS
  The depression test scores after DBS compared to baseline. Hamilton depression scale (HAMD, 0-64 scores, lower scores mean better outcome)

OTHER OUTCOMES:
Adverse Events Rate | 1 year and 3 years after DBS
  The rate of adverse events related to the implantation surgery or DBS devices.

CONTACTS AND LOCATIONS:
Overall Officials: Shuang Wang, MD, Principal Investigator — Epilepsy Center, Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- 2nd Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Fisher R, Salanova V, Witt T, Worth R, Henry T, Gross R, Oommen K, Osorio I, Nazzaro J, Labar D, Kaplitt M, Sperling M, Sandok E, Neal J, Handforth A, Stern J, DeSalles A, Chung S, Shetter A, Bergen D, Bakay R, Henderson J, French J, Baltuch G, Rosenfeld W, Youkilis A, Marks W, Garcia P, Barbaro N, Fountain N, Bazil C, Goodman R, McKhann G, Babu Krishnamurthy K, Papavassiliou S, Epstein C, Pollard J, Tonder L, Grebin J, Coffey R, Graves N; SANTE Study Group. Electrical stimulation of the anterior nucleus of thalamus for treatment of refractory epilepsy. Epilepsia. 2010 May;51(5):899-908. doi: 10.1111/j.1528-1167.2010.02536.x. Epub 2010 Mar 17. PMID 20331461
- [Result] Salanova V, Witt T, Worth R, Henry TR, Gross RE, Nazzaro JM, Labar D, Sperling MR, Sharan A, Sandok E, Handforth A, Stern JM, Chung S, Henderson JM, French J, Baltuch G, Rosenfeld WE, Garcia P, Barbaro NM, Fountain NB, Elias WJ, Goodman RR, Pollard JR, Troster AI, Irwin CP, Lambrecht K, Graves N, Fisher R; SANTE Study Group. Long-term efficacy and safety of thalamic stimulation for drug-resistant partial epilepsy. Neurology. 2015 Mar 10;84(10):1017-25. doi: 10.1212/WNL.0000000000001334. Epub 2015 Feb 6. PMID 25663221